CLINICAL TRIAL: NCT06778655
Title: Propolis in Management of Primary Herpetic Gingivostomatitis Measuring the Level of INF-γ in Saliva. Randomized Clinical Trial
Brief Title: Propolis in Primary Herpetic Gingivostomatitis
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Salsabeel A Afifi, PhD, lecturer of oral medicine and periodontology, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1212025
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Herpetic Gingivostomatitis
MeSH Terms: conditions — Stomatitis, Herpetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propolis group (Experimental)
  Interventions: Dietary Supplement: 5% propolis gel
- Control group (Placebo Comparator)
  Interventions: Other: Placebo gel

INTERVENTIONS:
Dietary Supplement: 5% propolis gel — 5% propolis gel (prepared according to Joshy et al. 2018) Joshy A, Doggalli N, Patil K, Kulkarni PK. To Evaluate the Efficacy of Topical Propolis in the Management of Symptomatic Oral Lichen Planus: A Randomized Controlled Trial. Contemp Clin Dent. 2018 Jan-Mar;9(1):65-71.
  Arms: Propolis group
Other: Placebo gel — placebo mucoadhesive gel having the same flavor, consistency, and color as the propolis.
  Arms: Control group

SUMMARY:
The purpose of the present study is to investigate the efficacy of 5% propolis gel in the treatment of primary herpetic gingivostomatitis in children and its effect on salivary IFN-γ levels.

ELIGIBILITY:
Inclusion Criteria:

* clinical manifestations suggestive of PHGS
* positive culture for HSV-1

Exclusion Criteria:

* negative culture for HSV-1
* allergic to honey or its products
* patients diagnosed with any systemic diseases, immunosuppressed or immunocompromised patients

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
The severity of oral lesions | one week
  mild, moderate, severe

SECONDARY OUTCOMES:
Pain | one week
  Visual Analogue Scale
measurement of salivary INF-γ level | one week
  by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Rania Shalaby, associate professor, Study Director — Fayoum University
Locations (1):
- fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Yes
upon request
Supporting Information: Study Protocol, SAP